CLINICAL TRIAL: NCT03379454
Title: The Impact of Melanoma and Drug Treatment in the Real World
Status: Completed | Type: Observational
Sponsor: Vitaccess Ltd (Industry)
Collaborators: Melanoma UK (Unknown); Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mark Larkin, Director, Vitaccess Ltd
Other Study IDs: 5100-01-2017
Record Dates: First submitted 2017-12-08; First posted 2017-12-20 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational, non-interventional registry study to collect real-world data from people living with melanoma and its treatment, which will be available to researchers to further the knowledge of melanoma and improve patient care.

DETAILED DESCRIPTION:
The registry uses Vitaccess' digital real-world evidence platform, and has been developed in collaboration with the patient advocacy group Melanoma UK.

Eligible participants install a study app on their smartphone or tablet. Researchers access aggregated, anonymised data via a cloud-based research portal. The platform provides benefits to participants, which it is hoped will encourage persistence with data submission; these include options to upload electronic documents such as scans, and access an online melanoma community.

The aggregated data are available in close to real time via "dashboards" and can be analysed according to a number of pre-set criteria (e.g. disease stage, age, geographic location).

State-of-the-art technologies and security policies are used in the platform to ensure industry-standard data storage and privacy for all users. Participants' personally identifiable information will remain confidential at all times, and researchers will not be able to identify individuals.

ELIGIBILITY:
Inclusion Criteria:

* adults with melanoma of any stage, resident in the UK with National Health Service (NHS) or Community Health Index (CHI) number, aged 18 and over, current or previous diagnosis of melanoma, willing to use their own smartphone or tablet.

Exclusion Criteria:

* no specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (age ≥18 years) with melanoma of any stage, who are resident in the UK, with NHS or CHI number, current or previous diagnosis of melanoma, willing to use their own smartphone or tablet.
Sampling Method: Non-Probability Sample
Enrollment: 819 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HRQL), general | Monthly throughout 4 year study duration
  EQ-5D-5L

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQL), oncology | Monthly throughout 4 year study duration
  QLQ-C30
Health-Related Quality of Life (HRQL), symptoms | Monthly throughout 4 year study duration
  PRO-CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Mark JW Larkin, PhD, Principal Investigator — Vitaccess Ltd
Locations (1):
- Vitaccess Ltd, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Aggregated data research dashboards will be available via industry subscriptions or free academic access.

REFERENCES:
- See also: Digital platform used to support the study — http://www.vitaccess.com
- See also: Research portal via which anonymised data can be made available to approved researchers — https://vitaccess.com/real-world-evidence/melanoma-uk-dataset/